CLINICAL TRIAL: NCT02866955
Title: Evaluation of the Efficacy of Estramustine in Patient With Breast Cancer Progression After Treatment With Aromatase Inhibitor.
Acronym: EFESE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-017788-40
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: aromatase inhibitors; Metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Estramustine; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP E (Estramustine) (Other): Patients with HER2-/RH+ breast cancer progressing after having already undergone a first line adjuvant treatment by estramustine
  Interventions: Drug: Estramustine
- GROUP T (Tamoxifen) (Other): Patients with HER2-/RH+ breast cancer progressing after having already undergone a first line adjuvant treatment by tamoxifen
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Estramustine — 140mg/4 caps/day
  Other Names: estramustine phosphate
  Arms: GROUP E (Estramustine)
Drug: Tamoxifen — 20mg/day
  Arms: GROUP T (Tamoxifen)

SUMMARY:
Despite advances in early detection and treatment strategy, about 25 to 40% of patients treated for breast cancer develop metastasis.

Some patients are in a therapeutic impasse situation. It is therefore necessary to consider all possible options. The Estramustine showed encouraging results in the treatment of metastatic breast cancer.

Given the clinical data, the answer rate of Estramustine and its impact on progression free survival deserve to be studied in earlier clinical situation.

This Phase II study evaluated the efficacy of Estramustine in women with breast cancer and metastates, already treated with aromatase inhibitors and for whom this treatment has failed.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women or women receiving Luteinizing hormone-releasing hormone (LHRH) analogs
* Histologically confirmed metastatic breast cancer RH+
* Measurable metastatic breast cancer (modified RECIST criteria) or not measurable but evaluable
* Recurrence:

  * being treated with aromatase inhibitors (AIs)
  * after adjuvant treatment by AIs
  * after progression of the metastatic cancer in patients receiving AIs following positive response during at least 6 months
* Performance status ≤ 2
* Haematological test: polynuclear neutrophiles ≥ 1.5 × 109 /L, haemoglobin ≥ 9 g/dL, blood platelet ≥ 100 × 109 /L
* Hepatic function: albumin ≥ 2.5 g/dL, serum bilirubin ≤ 1.5 × N (except if Gilbert's Syndrome) , aminotransferases ≤ 3 × N (≤ 5 × N if hepatic metastases)
* Renal function: serum creatinine ≤ 1.5 mg/dL or clearance of creatinine ≥ 40 ml/min
* Women without endometrial pathology
* Ability to provide written informed consent before the start of any study specific procedures

Exclusion Criteria:

* Age < 18 years old
* Pre-menopausal, pregnant or pregnant or breast feeding females
* Patient who should exclusively be treated by chemotherapy
* Women previously treated with chemotherapy but not by AIs
* Women previously treated by tamoxifen for their metastatic breast cancer
* HER2+
* Concurrent anti-cancer treatment (chemotherapy, surgery, immunotherapy, biological therapy and tumour embolism)
* Concurrent treatment with protocol-defined prohibited medications
* Malabsorption syndrome , significant digestive dysfunction, gastrectomy, jejunectomy, hemorrhagic recto colon
* Concurrent disease or condition that may interfere with study participation, or any serious medical disorder that would interfere with the subject's safety (for example, active or uncontrolled infection or any psychiatric condition prohibiting understanding or rendering of informed consent)
* Any pathology, including severe psychiatric or psychologic disease that may harm patient's safety or participation in the study
* Serious or not cured or unstable toxicity due to the administration of another drug being involved in clinical trials
* Uncontrolled cardiovascular pathologies
* Previous history of thromboembolic event like deep vein thrombosis or pulmonary embolism recorded within one year before the inclusion date
* Active uncontrolled infection
* Existence of an increased risk of thromboembolic event, apart from the metastatic cancer condition, such as:

  * known presence of antiphospholipid antibody
  * family history of thrombophilia
  * existence of any clinical, genetic, or biological abnormality which can increase the risk of thromboembolic event according to the
* Participation to a clinical trial at least 4 weeks prior the start of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06-15 (Actual); Primary Completion 2014-08-08 (Actual); Study Completion 2015-08-28 (Actual)

PRIMARY OUTCOMES:
Progression-free survival after a 6- month monotherapy with Estramustine in patients with HER2-/RH+ breast cancer progressing | up to 6 months
  proportion of patients in progression-free survival (PFS) after a 6-month treatment is defined as the duration of objective response or stabilisation of the disease according to the Recist criteria.
  The following events shall be considered as progressive :
  * Relapse
  * Treatment intolerance leading to stop the treatment
  * Death

SECONDARY OUTCOMES:
Risks of thrombosis | up to 6 months
  risks of thrombosis assessed by the analysis of biomarkers (D-Dimer, prothrombin fragment 1+2, von Willebrand factor, fibrinogen, Chain Reaction Protein)
Clinical benefit of estramustine | 1 year
  clinical benefit of estramustine assessed by RECIST criteria
Correlation between the answer rate and biomarkers | 1 year
  answer rate (RECIST criteria) and level of biomarkers (Lactate déshydrogénase, Antigène carcino-embryonnaire and Cancer antigène 15-3)
Tolerance of estramustine treatment | 1 year
  Toxicity (Common Terminology Criteria for Adverse Events)
Tolerance of tamoxifen treatments | 1 year
  Toxicity (Common Terminology Criteria for Adverse Events)
Proportion of patients developing thromboembolic events | 1 year
  proportion of patients developing thromboembolic events assessed in the 2 groups every month during the one-year patient follow-up

CONTACTS AND LOCATIONS:
Overall Officials: LUPORSI Elisabeth, MD, Principal Investigator — Institut de Cancérologie de Lorraine; GUASTALLA Jean Paul, MD, Principal Investigator — CLCC Léon Bérard
Locations (21):
- France (21):
  - Institut Sainte Catherine, Avignon
  - CHU Besançon-Jean Minjoz, Besançon
  - Polyclinique de Blois, Blois
  - CHU Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHRU Brest, Brest
  - Centre O. Lambret, Lille
  - CLCC Léon Bérard, Lyon
  - Hôpital Privé Clairval, Marseille
  - CHBM Site du Mittan, Montbéliard
  - CLCC Val d'Aurel, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Tenon, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Jean Godinot, Reims
  - Polyclinique Courlancy Reims, Reims
  - Clinique armoricaine, Saint-Brieuc
  - Centre Paul Strauss, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No